CLINICAL TRIAL: NCT00713037
Title: Hypoxia-PET and IMPT Dose Painting in Patients With Chordomas: A Pilot Study
Brief Title: Hypoxia-positron Emission Tomography (PET) and Intensity Modulated Proton Therapy (IMPT) Dose Painting in Patients With Chordomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tom DeLaney, MD, Attending Radiation Oncologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-162
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Chordoma
Keywords: fluoromisonidazole; PET scan; Hypoxia-PET; IMPT
MeSH Terms: conditions — Chordoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- (18F)-FMISO/CT (Experimental): The study utilizes PET/CT scanning with (18F)-FMISO/CT in addition to standard used CT and MRI. Patients enrolled in this trial completed 2 PET/CT investigations, the first before proton radiation therapy and the second at a dose of approximately 30 Gy (24-36 Gy).
  Interventions: Procedure: Fluoromisonidazole-PET/CT

INTERVENTIONS:
Procedure: Fluoromisonidazole-PET/CT — 2 scans at different time intervals: 2 weeks before and 3 weeks after the participants first proton radiation treatment.
  Other Names: FMISO-PET/CT

SUMMARY:
Before radiation treatment is given to treat chordomas, CT and MRI scans are used to create a three dimensional picture of the tumor using x-rays. The CT and MRI scans are used to determine the size and location of the area that will receive radiation treatment. The purpose of this research study is to see if combining the images from the FMISO-PET scan and the CT and MRI scans in radiation treatment planning changes the size and location of the area that will receive radiation treatment when compared to planning the radiation treatment with CT and MRI scans alone.

DETAILED DESCRIPTION:
* In this research study we are determining whether the positron emission tomography (PET) investigation performed with the investigational radioactive substance FMISO can show areas of tumor with lower oxygen levels. There is evidence that tumor with low oxygen levels are more resistant to radiation therapy. CT and MRI scans are not able to detect these oxygen levels in tumors.
* Participants will be asked to have the FMISO-PET/CT scan at 2 different times. It will be performed 2 weeks before and 3 weeks after the participants first proton radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Skull base and spinal chordomas diagnosis based on pathology review by Department of Pathology at Massachusetts General Hospital
* Patient to be treated with proton or combined photon RT for primary CD or recurrent CD after surgery
* 18 years of age or older
* Karnofsky Score of 60% or greater
* Gross tumor mass larger than 1cm (maximal diameter on MRI)

Exclusion Criteria:

* Recurrences after RT
* Pregnancy
* Allergic reaction to FMISO injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To evaluate if FMISO-PET is a feasible approach for the visualization of hypoxia in skull base and spinal CD. | 2 years

SECONDARY OUTCOMES:
To investigate if using a Dose Painting/IMPT approach based on FMISO-PET/CT/MRI the irradiation dose can be escalated and the normal tissue be better spared in comparison to a IMPT approach based on anatomical imaging alone. | 2 years
To evaluate and improve the precision of patients' positioning and image fusin using PET/CT for radiation treatment planning. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F. DeLaney, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States